CLINICAL TRIAL: NCT04427007
Title: Moisture Management Liner Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Vivonics, Inc. (Industry)
Responsible Party: Principal Investigator, Todd Farrell, Director of Research, Liberating Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: E00572.1a; 2020/01/1 (Other: Solutions IRB)
Record Dates: First submitted 2020-05-26; First posted 2020-06-11 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Amputation Stumps; Amputees; Amputation; Lower Limb Deformities, Congenital; Prosthesis User; Prosthesis
Keywords: cooling; amputee; lower limb difference; Prosthetic; socket; Prosthesis; Prosthetist; Liner; sweat; walking; sock; leg; perspiration; moisture; heat; thermal
MeSH Terms: conditions — Lower Extremity Deformities, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Prosthetic Liner (Experimental): Participants will test the experimental prosthetic liner by walking on a treadmill while wearing the liner.
  Interventions: Device: Moisture Management Liner
- Control Prosthetic Liner (Other): Participants will test the control (participant's usual) liner by walking on a treadmill while wearing the liner.
  Interventions: Device: Control Liner

INTERVENTIONS:
Device: Moisture Management Liner — A prototype prosthetic liner designed to reduce and/or remove moisture and heat that builds up on the limb.
  Arms: Experimental Prosthetic Liner
Device: Control Liner — The participant's usual prosthetic liner
  Arms: Control Prosthetic Liner

SUMMARY:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by non-breathable and non- thermally conductive materials that can create a warm and ultimately moist environment.

The investigators have developed a silicone liner approach to remove sweat from the skin and out of the socket and to passively conduct heat from the skin using thermally conductive elastomers. This liner has been developed to work alongside a thermo-electric cooling (TEC)-based module called the Intrasocket Cooling Element (ICE) developed in a parallel project by Vivonics, Inc. and Liberating Technologies, Inc. The ICE device can be embedded into the prosthesis in order to cool the residual limb. A technology that can provide thermal control while retaining adequate suspension, weight, and other prosthetic characteristics would benefit many prosthesis wearers.

DETAILED DESCRIPTION:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by non-breathable and non- thermally conductive materials that can create a warm and ultimately moist environment. These layers consist of a prosthetic liner that rolls onto the limb and traps heat and occasional extra prosthetic socks. Studies found increases in socket temperature after the prosthesis was donned. Temperatures were found to remain elevated long after activity cessation and even a rest period of double the duration of the preceding activity period is insufficient to return the limb to its initial temperature. A small amount of activity can cause the socket temperature to elevate and remain at an uncomfortable level for an extended period of time, which can lead to decreased wear times. In summary, an uncomfortable socket/residual limb interface decreases prosthesis use among amputees who want to remain active in their lives.

To address this, the investigators have developed a silicone liner approach to remove sweat from the skin and out of the socket and to passively conduct heat from the skin using thermally conductive elastomers. This liner has been developed to work alongside a thermo-electric cooling (TEC)-based module called the Intrasocket Cooling Element (ICE) developed in a parallel project by Vivonics, Inc. and Liberating Technologies, Inc. The ICE device can be embedded into the prosthesis in order to cool the residual limb. A technology that can provide thermal control while retaining adequate suspension, weight, and other prosthetic characteristics would benefit many prosthesis wearers.

This study will focus on investigating the efficacy of this novel moisture and thermal management (experimental) liner.

The rationale for this study is to determine how well the new technology can regulate the residual limb temperature, reduce the moisture generation, and remove excess moisture in a controlled laboratory environment.

The objective of this study is to measure the effects experimental techniques of moisture and thermal management has on moisture and temperature in the socket. Moisture and thermal management of the residual limb inside the prosthetic socket could result in greater comfort while wearing the prosthesis, and ultimately could result in greater function and better quality of life (QoL). Other measures that may be collected are exploratory.

A repeated measures study will be conducted to analyze the temperature and moisture generation of the residual limb with and without the experimental liner and active cooling system within a standard prosthetic socket.

Both able-bodied research subjects, and lower limb amputee research subjects who use transfemoral or transtibial prostheses will be recruited for testing. Liners for able-bodies subjects will have the distal end removed to allow for donning. All subjects will visit Liberating Technologies, Inc. to be consented and to complete study testing.

A maximum of 10 able-bodied and 20 lower-limb amputee subjects will be recruited for this study. This is increased from a target 12 subjects to account for any drop-outs, etc.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputee
* Be willing and able to complete the tasks outlined
* Are at least 6 months on a definitive prosthesis
* Fits within an experimental liner
* Can understand English in order to be properly consented and provide their feedback to the study personnel

Exclusion Criteria:

* The risks to pregnant women and fetuses are unknown and therefore pregnant women should not participate in the study
* Other unforeseen disqualifying criteria (such as specific cognitive issues, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2022-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Liberating Technologies, Inc., Holliston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Liner, Then Control Liner: Participants will test the experimental prosthetic liner by walking on a treadmill while wearing the liner. They will then test the control liner by walking on the treadmill while wearing their usual prosthetic liner.
  Moisture Management Liner: A prototype prosthetic liner designed to reduce and/or remove moisture and heat that builds up on the limb.
- Control Liner, Then Experimental Liner: Participants will test the control (participant's usual) liner by walking on a treadmill while wearing the liner. They will then test the experimental prosthetic liner by walking on a treadmill while wearing the liner.
  Control Liner: The participant's usual prosthetic liner
Period: Overall Study
Arm/Group | Experimental Liner, Then Control Liner | Control Liner, Then Experimental Liner
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Unable to use the experimental liner due to suspension issues. Incomplete data collection. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Liner, Then Control Liner | Control Liner, Then Experimental Liner | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Residual Limb Temperature
Description: Changes in residual limb temperature during walking/resting measured with temperature sensors placed on the limb. Positive values signify a raise in temperature and negative values signify a drop in temperature between the start of walking to the end of walking.
Time Frame: 2 hours
Population: Data only reported for the subject who completed both conditions.
Measure: Number; unit: Degrees Fahrenheit
Arm/Group | Experimental Prosthetic Liner | Control Prosthetic Liner
Number analyzed (Participants) | 1 | 1
Degrees Fahrenheit | 3.0 | 3.2

ADVERSE EVENTS:
Time Frame: During the in-lab visit (about 2-4 hours)
Arm/Group | Experimental Prosthetic Liner | Control Prosthetic Liner
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04427007/Prot_001.pdf